CLINICAL TRIAL: NCT02710747
Title: The Pharmacogenetics of Optimal Warfarin Therapy in Chinese Patients After Heart Valve Replacement.
Acronym: POWAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDREC2014265H
Record Dates: First submitted 2016-02-25; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2015-12

CONDITIONS: Heart Valve Disease; Older Than 18-years-old; Without Any Liver or Kidney Diseases
Keywords: warfarin; Chinese patients; heart valve replacement
MeSH Terms: conditions — Heart Valve Diseases; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genetic Group (Experimental): Dose (mg/week) = [5.6044 - 0.02614 × Age [in years] + 0.0087 × Height [cm] + 0.0128 × Weight [kg] - 0.8677 × VKORC1 A/G -1.6974 × VKORC1 A/A - 0.5211 × CYP2C9 *1/*2 - 0.9357 × CYP2C9 *1/*3 - 1.0616 × CYP2C9 *2/*2 - 1.9206 × CYP2C9*2/*3 - 2.3312 × CYP2C9 *3/*3 - 0.1092 × Asian race - 0.5503 × amiodarone ]2
  Interventions: Genetic: CYP2C9;VKORC1
- Control Group (No Intervention): Dose for the first three days after operation will be 4.5mg/d.

INTERVENTIONS:
Genetic: CYP2C9;VKORC1
  Arms: Genetic Group

SUMMARY:
To value the accuracy of the dosing algorithm published by the International Warfarin Pharmacogenetics Consortium in Chinese patients after heart valve replacement.

To value the accuracy of warfarin pharmacogenomics algorithm by the algorithm calculated dose and actual dose in the Chinese patients.

DETAILED DESCRIPTION:
The dosing algorithm published by the International Warfarin Pharmacogenetics Consortium hadn't been verifying by a standard randomized prospective study in Chinese patients after heart valve replacement. And, warfarin will affect people's coagulation, so that probably increase the drainage. We'll analyse the interaction of patients' PT-INR or drainge and oral warfarin dosing.

ELIGIBILITY:
Inclusion Criteria:atrial fibrillation

* atrial fibrillation
* heart valve replacement
* VTE

Exclusion Criteria:

* severe liver or kidney diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The perccentage of time that the INR was in the therapeutic range | 3 months

SECONDARY OUTCOMES:
all drainage fluid of every patient | 1 week after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China